CLINICAL TRIAL: NCT04897230
Title: The Effects of Acute Yoga Practice on Heart Rate and Heart Rate Variability Responses to Mental Stress
Brief Title: Effects of Yoga on Heart Rate and Heart Rate Variability Responses to Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KMUH-IRB-20120375
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Reactivity to Stress
Keywords: yoga, mental stress, cardiac autonomic function, stress response
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga Condition (Active Comparator): An experienced yoga instructor led the 30 minutes yoga condition session which consisted of 5 minutes warm up, 5 minutes breathing exercises, and 20 minutes yoga poses practice. The yoga props were used according to each participant's particular body type and needs to help he/she achieve precise yoga postures safely and comfortably.
  Interventions: Behavioral: Hatha Yoga
- Control Condition (Placebo Comparator): Participants in the control condition were watching a neutral video on a television.
  Interventions: Behavioral: Video Watching

INTERVENTIONS:
Behavioral: Hatha Yoga — The yoga poses were chosen for providing a restorative session based on their purported relationship to restorative effects to best promote cardiac autonomic recovery from mental stress.
  Arms: Hatha Yoga Condition
Behavioral: Video Watching — The video was about the history of the Earth which encompasses the development of the planet Earth from its formation to the present day.
  Arms: Control Condition

SUMMARY:
Introduction: Yoga has been shown to reduce stress and have benefits for a number of stress-related disorders. However, the effects of an acute bout of yoga practice on cardiac autonomic response to and recovery from stress remain unclear. This study aimed to examine the effect of a single bout of yoga on heart rate (HR) and heart rate variability (HRV) response to and recovery from mental stress.

Materials and Methods: This study was conducted with a randomized, counterbalanced, crossover design. A total of 44 participants completed two sessions (yoga and video watching (VW)) in randomly assigned order. After each condition, participants underwent a Stroop task and mental arithmetic task. Electrocardiogram was measured and HR and HRV for resting, each condition, and the stress and recovery periods were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 40 years old
* a body mass index (BMI) between 18.5 and 30
* being sedentary

Exclusion Criteria:

* Electrocardiogram (ECG) abnormalities (e.g., arrhythmia, atrioventricular blocks)
* history of cardiovascular disease, diabetes, or renal disease
* contraindications for exercise (e.g., orthopedic problems)
* involvement in any yoga practice
* being pregnant or nursing
* use of tobacco products or medications that may affect cardiovascular function

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate | up to 5 minutes
  Heart rate was derived from continuous heart rate recording, at a sampling rate of 1024 Hz, using an electrocardiogram (ECG) system
Heart Rate Variability | up to 5 minutes
  Heart rate variability was derived from continuous heart rate recording, at a sampling rate of 1024 Hz, using an electrocardiogram (ECG) system

IPD SHARING:
Plan to Share IPD: No